CLINICAL TRIAL: NCT07103408
Title: A Phase II Study Evaluating Concurrent Chemoradiotherapy Combined With Dual Immune Checkpoint Blockade (PD-1/CTLA-4) for Limited-stage Small Cell Lung Cancer
Brief Title: A Study Evaluating Concurrent Chemoradiotherapy Combined With Dual Immune Checkpoint Blockade for Limited-stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10136
Record Dates: First submitted 2025-07-16; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Small-Cell Lung Cancer (SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study group (Experimental): Patients will receive chemotherapy (etoposide and platinum-based drugs) combined with dual immune checkpoint blockade (iparomlimab and tuvonralimab) and thymosin alpha 1, with a total cycles of 4. Thoracic radiotherapy was performed no later than the three cycle of chemotherapy. Prophylactic cranial irradiation was recommended for patients who received complete response or partial response after chemoradiotherapy. Finally consolidation therapy with dual immune checkpoint blockade (iparomlimab and tuvonralimab) and thymosin alpha 1 was conducted for one year.
  Interventions: Drug: Immuno-chemotherapy; Radiation: Radiotherapy; Drug: Consolidative therapy

INTERVENTIONS:
Drug: Immuno-chemotherapy — Immuno-chemotherapy regimen included etoposide, cisplatin, iparomlimab and tuvonralimab, and thymosin alpha 1.
Radiation: Radiotherapy — Definitive dose of thoracic radiotherapy was delivered no later than the three cycle of immuno-chemotherapy.
  Prophylactic cranial irradiation (PCI) was delivered with a total dose of 25Gy in 10 fractions. PCI was recommended for patients who achieved complete response or partial response after thoracic chemoradiotherapy.
Drug: Consolidative therapy — Consolidation therapy regimen included iparomlimab and tuvonralimab, and thymosin alpha 1, with a duration of one year.

SUMMARY:
This study will enroll patients with limited-stage small cell lung cancer (SCLC). Patients will receive chemotherapy (etoposide and platinum-based drugs) combined with dual immune checkpoint blockade (PD-1/CTLA-4) and thymosin alpha 1, with a total cycles of 4. Thoracic radiotherapy was performed no later than the three cycle of chemotherapy. Prophylactic cranial irradiation was recommended for patients who received complete response or partial response after chemoradiotherapy. Finally consolidation therapy with dual immune checkpoint blockade (PD-1/CTLA-4) and thymosin alpha 1 was conducted for one year. The study aims to evaluate the efficacy and safety of this treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 75 years or older;
* Patients must have histologically or cytologically confirmed small cell lung cancer (SCLC);
* Stage II-III according to AJCC 8th staging system;
* No prior chemotherapy, radiotherapy, surgery, targeted therapy, or immunotherapy;
* Expected survival ≥ 12 weeks;
* WHO Performance Status (PS) score of 0 or 1;
* Female subjects must not be breastfeeding;
* Women of childbearing potential (WOCBP) must agree to use contraception during the study treatment and for 5 months after the last dose of study drug (i.e., 30 days [one ovulation cycle] plus approximately five half-lives of the study drug);
* Adequate organ and bone marrow function as defined by the following criteria:
* Forced Expiratory Volume in 1 second (FEV1) ≥ 800 mL;
* Absolute neutrophil count ≥ 1.5 × 10⁹/L;
* Platelets ≥ 100 × 10⁹/L;
* Hemoglobin ≥ 9.0 g/dL;
* Creatinine clearance ≥ 50 mL/min as calculated by the Cockcroft-Gault formula (Cockcroft and Gault, 1976);
* Serum bilirubin ≤ 1.5 × upper limit of normal (ULN);
* AST and ALT ≤ 2.5 × ULN.

Exclusion Criteria:

* Concurrent enrolment in another clinical study, unless it is an observational(non-interventional) clinical study;
* Mixed small cell and non-small cell lung cancer histology;
* Prior use of anti-PD-1, anti-PD-L1, or anti-CTLA4 antibodies;
* Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access;
* Active or prior documented autoimmune disease within the past 2 years;
* Active or prior documented inflammatory bowel disease (eg. Crohn's disease, ulcerative colitis);
* History of primary immunodeficiency;
* History of organ transplant that requires therapeutic immunosuppression;
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent;
* Known history of tuberculosis;
* History of another primary malignancy within 5 years prior to starting treatment, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and the disease under study;
* Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2-year
  PFS measures the time from the start date of treatment to disease progression, death from any cause or last follow up if alive.

SECONDARY OUTCOMES:
Overall survival | 2-year
  OS measures the time from the start date of treatment to death from any cause or last follow up if alive.
Treatment-related toxicity | through study completion, an average of 18 months
  Treatment-related toxicities were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) 5.0 toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garaci E, Pica F, Serafino A, Balestrieri E, Matteucci C, Moroni G, Sorrentino R, Zonfrillo M, Pierimarchi P, Sinibaldi-Vallebona P. Thymosin alpha1 and cancer: action on immune effector and tumor target cells. Ann N Y Acad Sci. 2012 Oct;1269:26-33. doi: 10.1111/j.1749-6632.2012.06697.x. PMID 23045967
- [Background] Malhotra J, Chiappori A, Fujioka N, Hanna NH, Feldman LE, Patel M, Moore D, Chen C, Jabbour SK. Phase I/II trial of plinabulin in combination with nivolumab and ipilimumab in patients with recurrent small cell lung cancer (SCLC): Big ten cancer research consortium (BTCRC-LUN17-127) study. Lung Cancer. 2024 Sep;195:107932. doi: 10.1016/j.lungcan.2024.107932. Epub 2024 Aug 21. PMID 39173229
- [Background] Huang Y, Yang Y, Zhao Y, Zhao H, Zhou N, Zhang Y, Chen L, Zhou T, Chen G, Wu T, Lu L, Xue S, Kang X, Zhang L, Fang W. QL1706 (anti-PD-1 IgG4/CTLA-4 antibody) plus chemotherapy with or without bevacizumab in advanced non-small cell lung cancer: a multi-cohort, phase II study. Signal Transduct Target Ther. 2024 Jan 29;9(1):23. doi: 10.1038/s41392-023-01731-x. PMID 38282003
- [Background] Cheng W, Kang K, Zhao A, Wu Y. Dual blockade immunotherapy targeting PD-1/PD-L1 and CTLA-4 in lung cancer. J Hematol Oncol. 2024 Jul 27;17(1):54. doi: 10.1186/s13045-024-01581-2. PMID 39068460
- [Background] Duan H, Shi L, Shao C, Wang Y, Wang Z, Ni Y, Zhao J, Sun J, Tong L, Lei J, Jiang T, Liu Z, Yan X. A multicenter, single-arm, open study of neoadjuvant or conversion atezolizumab in combination with chemotherapy in resectable small cell lung cancer (Cohort Study). Int J Surg. 2023 Sep 1;109(9):2641-2649. doi: 10.1097/JS9.0000000000000501. PMID 37428211
- [Background] Cheng Y, Spigel DR, Cho BC, Laktionov KK, Fang J, Chen Y, Zenke Y, Lee KH, Wang Q, Navarro A, Bernabe R, Buchmeier EL, Chang JW, Shiraishi Y, Sezgin Goksu S, Badzio A, Shi A, Daniel DB, Hoa NTT, Zemanova M, Mann H, Gowda H, Jiang H, Senan S; ADRIATIC Investigators. Durvalumab after Chemoradiotherapy in Limited-Stage Small-Cell Lung Cancer. N Engl J Med. 2024 Oct 10;391(14):1313-1327. doi: 10.1056/NEJMoa2404873. Epub 2024 Sep 13. PMID 39268857